CLINICAL TRIAL: NCT00863811
Title: Effects of the Oral Administration of an Association of Forskolin With Rutin and Vitamins B on Intraocular Pressure in Patients Affected by Primary Open Angle Glaucoma and Treated With Either Beta-blockers or Prostaglandin Eye Drops
Brief Title: Effects of Forskolin on Intraocular Pressure in Glaucomatous Patients Under Treatment With Either Beta-blockers or Prostaglandins Eye Drops
Status: Withdrawn | Type: Observational
Why Stopped: loss of interest before enrolment started
Sponsor: Sooft Italia (Industry)
Responsible Party: Michele Vetrugno, Ophthalmology Dept., University of Bari, Italy
Other Study IDs: KRONEK-PG-BB
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Primary Open Angle Glaucoma; Intraocular Pressure
Keywords: POAG; IOP; Forskolin; beta-blockers; prostaglandins
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 2: POAG patients with IOP under control by prostaglandins eye drops treatment and assuming two tablets per day of the food supplement KRONEK
- 1: POAG patients compensated by the treatment of betablockers eye drops and taking two tablets per day of KRONEK

SUMMARY:
Elevated intraocular pressure is still the main risk factor for development and progression of glaucoma. Several drugs exist on the market that may decrease IOP in glaucomatous patients. However, some patients cannot reach the target pressure despite a multitherapy with a combination of drugs, and are therefore addressed to surgical treatments. Forskolin is a natural compound that is a receptor-independent adenyl-cyclase activator, that increases intracellular cAMP. It has been shown to be able to decrease IOP after topical application, by a mechanism that is not used by the other drugs. Aim of the present study is to see whether oral administration of a food supplement containing forskolin (KRONEK) has any effect on the IOP of POAG patients with stable IOP obtained by treatment with either beta-blockers or prostaglandins.

ELIGIBILITY:
Inclusion Criteria:

* Primary Open Angle Glaucoma associated with ocular hypertension
* Target pressure achieved by single-agent therapy (beta-blockers or prostaglandins)
* Visual acuity > 6/10

Exclusion Criteria:

* Miopy or Hypermetropy > 5D
* Concomitant ocular pathologies
* Previous ocular surgery
* Known hypersensitivity to any of the components in the KRONEK tablets
* Concomitant participation in other trials
* Changes of topic glaucoma therapy during the course of the study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by POAG and already under observation in the centers that take part in this study
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure | Enrollment, 1, 2, 3 months

SECONDARY OUTCOMES:
Intraocular pressure fluctuations during the day | Enrollment, 1, 2, 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Michele Vetrugno, MD, Principal Investigator — Ophthalmology Department, University of Bari
Locations (1):
- Ophthalmology Department of the University, Bari, Italy

REFERENCES:
- [Background] Caprioli J, Sears M. Forskolin lowers intraocular pressure in rabbits, monkeys, and man. Lancet. 1983 Apr 30;1(8331):958-60. doi: 10.1016/s0140-6736(83)92084-6. PMID 6132271
- [Background] Caprioli J, Sears M. The adenylate cyclase receptor complex and aqueous humor formation. Yale J Biol Med. 1984 May-Jun;57(3):283-300. PMID 6093393
- [Background] Lee PY, Podos SM, Howard-Williams JR, Severin CH, Rose AD, Siegel MJ. Pharmacological testing in the laser-induced monkey glaucoma model. Curr Eye Res. 1985 Jul;4(7):775-81. doi: 10.3109/02713688509020033. PMID 3861296